CLINICAL TRIAL: NCT03621735
Title: Reversing Synchronized Brain Circuits With Targeted Auditory-Somatosensory Stimulation to Treat Phantom Percepts- Stage 2
Brief Title: Reversing Synchronized Brain Circuits With Targeted Auditory-Somatosensory Stimulation to Treat Phantom Percepts
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Susan E. Shore, Professor, Otolaryngology, Molecular and Integrative Physiology; Professor, Biomedical Engineering Kresge Hearing Research Institute The Joseph Hawkins Collegiate Research Professor, University of Michigan
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HUM00143675; 1RF1MH114244 (NIH)
Record Dates: First submitted 2018-07-30; First posted 2018-08-08 (Actual); Results first posted 2023-08-30 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Tinnitus
Keywords: Tinnitus; Ringing in the ear
MeSH Terms: conditions — Tinnitus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Sham then Active (Other): Active: Bimodal auditory-somatosensory stimulation
  Sham: Sham Bimodal auditory-somatosensory stimulation
  Subjects receive both a sham treatment and an active treatment. The subjects will be blinded to which treatment they are receiving. Both treatments are delivered using a take-home device programmed in the lab.
  During active treatment, the device will deliver electric somatosensory and auditory stimulation.
  Interventions: Device: Burst-SCS/sham SCS
- Active then Sham (Other): Active: Bimodal auditory-somatosensory stimulation
  Sham: Sham Bimodal auditory-somatosensory stimulation
  Subjects receive both an active treatment and a sham treatment. The subjects will be blinded to which treatment they are receiving. Both treatments are delivered using a take-home device programmed in the lab.
  During active treatment, the device will deliver electric somatosensory and auditory stimulation.
  Interventions: Device: Sham SCS/Burst-SCS

INTERVENTIONS:
Device: Burst-SCS/sham SCS — The auditory stimulus will be individualized based on subject baseline audiogram and tinnitus test results and is presented through a calibrated earphone.
  Somatosensory stimulation will be delivered by pads positioned on the cheek overlying the trigeminal ganglion or on the neck at overlying cervical nerves, c1 or c2, determined by the manner in which the subject can modulate the tinnitus.
  For each arm of the study subjects will have daily treatments for 30-60 minutes for 6 weeks.
  Other Names: St. Jude Medical Invisible Trial System
  Arms: Sham then Active
Device: Sham SCS/Burst-SCS — Somatosensory stimulation will be delivered by pads positioned on the cheek overlying the trigeminal ganglion or on the neck at overlying cervical nerves, c1 or c2, determined by the manner in which the subject can modulate the tinnitus.
  The auditory stimulus will be individualized based on subject baseline audiogram and tinnitus test results and is presented through a calibrated earphone.
  For each arm of the study subjects will have daily treatments for 30-60 minutes for 6 weeks.
  Other Names: St. Jude Medical Invisible Trial System
  Arms: Active then Sham

SUMMARY:
The goal of the study is to reduce tinnitus (ringing in the ear) loudness and improve the quality of life for those that are affected by tinnitus. This study will enroll subjects who have constant and bothersome tinnitus with no greater than a mild hearing loss up to 6 kHz, and no greater than a moderate hearing loss in the tinnitus frequencies. Subjects must also have the ability to alter the loudness or pitch of the ringing in their ears by performing a head, neck, face, or upper body movement. Subjects will be given both the treatment and sham arms (the study will randomly assign which arm is administered first) and will have a washout period of 6 weeks after each arm. The study will take approximately 36 weeks for subjects to complete and will enroll up to 300 individuals.

ELIGIBILITY:
Inclusion Criteria:

* Must report constant, subjective, preferably unilateral tinnitus without any active external or middle ear pathology.
* No greater than a mild hearing loss up to 6 kHz, and no greater than a moderate hearing loss at the tinnitus frequencies.
* Must be able to modulate their tinnitus with a somatic maneuver
* Preferably onset of tinnitus less than one year ago, but present for at least 6 months. Tinnitus should be bothersome.
* Absence of retrocochlear pathology/8th nerve lesion
* No participation in a tinnitus treatment regimen within the past six months or participation in the University of Michigan stage 1 clinical trial.

Exclusion Criteria:

* Diagnosis of Meniere's disease
* Diagnosis of Semicircular Canal Dehiscence
* Unilateral or bilateral cochlear implant recipients
* Diagnosis of acoustic neuroma
* Evidence of retrocochlear disease
* Certain medications and conditions (will be reviewed at screening)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2022-07-06 (Actual); Study Completion 2022-07-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Shore, Ph.D., Principal Investigator — University of Michigan
Locations (1):
- The University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jones GR, Martel DT, Riffle TL, Errickson J, Souter JR, Basura GJ, Stucken E, Schvartz-Leyzac KC, Shore SE. Reversing Synchronized Brain Circuits Using Targeted Auditory-Somatosensory Stimulation to Treat Phantom Percepts: A Randomized Clinical Trial. JAMA Netw Open. 2023 Jun 1;6(6):e2315914. doi: 10.1001/jamanetworkopen.2023.15914. PMID 37266943

RESULTS

PARTICIPANT FLOW:
Groups:
- Active Then Sham: Active: Bimodal auditory-somatosensory stimulation
  Sham: Sham Bimodal auditory-somatosensory stimulation
  Subjects receive both an active treatment and a sham treatment. The subjects will be blinded to which treatment they are receiving. Both treatments are delivered using a take-home device programmed in the lab.
  During active treatment, the device will deliver electric somatosensory and auditory stimulation.
  Sham SCS/Burst-SCS: Somatosensory stimulation will be delivered by pads positioned on the cheek overlying the trigeminal ganglion or on the neck at overlying cervical nerves, c1 or c2, determined by the manner in which the subject can modulate the tinnitus.
  The auditory stimulus will be individualized based on subject baseline audiogram and tinnitus test results and is presented through a calibrated earphone.
  For each arm of the study subjects will have daily treatments for 30-60 minutes for 6 weeks.
- Sham Then Active: Active: Bimodal auditory-somatosensory stimulation
  Sham: Sham Bimodal auditory-somatosensory stimulation
  Subjects receive both a sham treatment and an active treatment. The subjects will be blinded to which treatment they are receiving. Both treatments are delivered using a take-home device programmed in the lab.
  During active treatment, the device will deliver electric somatosensory and auditory stimulation.
  Burst-SCS/sham SCS: The auditory stimulus will be individualized based on subject baseline audiogram and tinnitus test results and is presented through a calibrated earphone.
  Somatosensory stimulation will be delivered by pads positioned on the cheek overlying the trigeminal ganglion or on the neck at overlying cervical nerves, c1 or c2, determined by the manner in which the subject can modulate the tinnitus.
  For each arm of the study subjects will have daily treatments for 30-60 minutes for 6 weeks.
Period: Overall Study
Arm/Group | Active Then Sham | Sham Then Active
Started | 50 | 50
Received Device or Sham Device to Use | 49 | 50
Began First Washout Period | 41 | 44
Began Crossover Assignment | 39 | 40
Began Second Washout Period | 39 | 39
Began 12-Week Follow Up | 38 | 39
Completed | 37 | 37
Not Completed | 13 | 13
Not completed — Withdrawal by Subject | 13 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Then Sham | Sham Then Active | Total
Number analyzed (Participants) | 49 | 50 | 99
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.0 (1.8) | 47.1 (1.8) | 47.1 (1.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 22 | 39
  Male | 32 | 28 | 60
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 48 | 48 | 96
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 5 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 44 | 45 | 89
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 49 | 50 | 99
Objective Tinnitus Loudness [Mean (Standard Deviation); unit: decibels] — Participants are guided through a self-directed computerized assessment software (TinnTester) that estimates how loud (in decibels) they perceive their tinnitus to be.
  decibels | 57.0 (13.7) | 55.1 (13.4) | 56.1 (13.5)
Tinnitus Functional Index (TFI) [Mean (Standard Deviation); unit: score on a scale] — TFI is a clinical questionnaire that assesses tinnitus impact on a subject's quality of life. It uses a scale of 0 - 100 where 0 means no negative impact on quality of life from tinnitus and 100 is devastating impact.
  score on a scale | 43.1 (13.4) | 42.6 (16.8) | 42.9 (15.1)
Tinnitus Handicap Inventory (THI) [Mean (Standard Deviation); unit: score on a scale] — A 25-item questionnaire which assesses subjective impacts of tinnitus related to quality of life on a 100-point numeric scale. Scores 17 points or higher are considered bothersome tinnitus. The higher scores reflecting greater self-perceived tinnitus handicap.
  score on a scale | 37.9 (17.7) | 34.9 (18.3) | 36.4 (18)
Minimum Masking Level (MML) [Mean (Standard Deviation); unit: dB (sensation level)] | 35.4 (12.9) | 33.0 (12.2) | 34.2 (12.6)
Tinnitus Hearing Survey [Mean (Standard Deviation); unit: score on a scale] — 10-question survey with a scale from 0 to 4 to determine if active treatment has an effect or interaction with perceived handicap due to hearing loss and sound level tolerance. Categories are comprised of tinnitus, hearing, and sound tolerance. An answer of 0 is no/not a problem, and an answer of 4 is yes/a very big problem.
  score on a scale | 5.9 (2.5) | 5.2 (3) | 5.6 (2.8)

OUTCOME MEASURES:

1. Primary Outcome: Change in Objective Tinnitus Loudness
Description: Change in Tinnitus by the TinnTester software. Participants are guided through a self-directed computerized assessment software that estimates how loud (in decibels) they perceive their tinnitus to be (TinnTester). These will be collected weekly during each treatment arm and washout. Absolute differences are averaged relative to baseline to determine loudness change.
  For each of the two arms, Active Then Sham and Sham Then Active, data is presented at the end of each arm phase group, in six week intervals. Thus Active First below is at 6 weeks after baseline, Washout is at 12 weeks, Active First then Sham at 18, and Active First then Sham Washout at 24 and the same pattern for the Sham First group.
Time Frame: Up to 24 weeks
Population: Because of the crossover nature of this trial, and to determine whether spillover effects were present, participants are represented multiple times for each segment of the trial in which they participated.
Measure: Mean (Standard Error); unit: decibels sensation level (dB SL)
Groups:
- Active First: Participants who were assigned to the bimodal auditory-somatosensory stimulation (intervention) initially following randomization and completed treatment.
- Active-First Washout: Participants who received the intervention initially following randomization and completed the first washout period.
- Active-First Then Sham: Participants who initially received the intervention following randomization and completed treatment with the sham bimodal auditory-somatosensory stimulation (sham) following the first washout period.
- Active-First-Then-Sham Washout: Participants who completed the second washout after initially receiving the intervention following randomization and then received the sham following the first washout period.
- Sham First: Participants who were assigned to the sham bimodal auditory-somatosensory stimulation (sham) initially following randomization and completed treatment.
- Sham-First Washout: Participants who received the sham initially following randomization and completed the first washout period.
- Sham-First Then Active: Participants who initially received the sham following randomization and completed treatment with the bimodal auditory-somatosensory stimulation (intervention) following the first washout period.
- Sham-First-Then-Active Washout: Participants who completed the second washout after initially receiving the sham following randomization and then received the intervention following the first washout period.
Arm/Group | Active First | Active-First Washout | Active-First Then Sham | Active-First-Then-Sham Washout | Sham First | Sham-First Washout | Sham-First Then Active | Sham-First-Then-Active Washout
Number analyzed (Participants) | 41 | 40 | 39 | 39 | 44 | 40 | 39 | 38
decibels sensation level (dB SL) | -6.1 (1.8) | -9.5 (2.1) | -10.2 (2.3) | -11.0 (2.5) | -3.7 (1.3) | -4.7 (1.5) | -5.8 (2.3) | -4.9 (2.4)

2. Primary Outcome: Change in Tinnitus Functional Index (TFI)
Description: TFI is a clinical questionnaire that assesses tinnitus impact on a participant's quality of life. It uses a scale of 0 - 100 where 0 means no negative impact on quality of life from tinnitus and 100 is devastating impact. These will be collected weekly during each treatment arm and washout.
  For each of the two arms, Active Then Sham and Sham Then Active, data is presented at the end of each arm phase group, in six week intervals. Thus Active First below is at 6 weeks after baseline, Washout is at 12 weeks, Active First then Sham at 18, and Active First then Sham Washout at 24 and PSM 36 weeks, and the same pattern for the Sham First group. Values presented are all shown as change from baseline.
Time Frame: Up to 36 weeks
Measure: Mean (Standard Error); unit: Points on a Scale
Groups:
- Active-First Post-Study Monitoring (PSM) Period: Participants who received the intervention initially following randomization, and who completed the follow-up period.
- Sham-First Post-Study Monitoring (PSM) Period: Participants who received the sham initially following randomization, and who completed the follow-up period.
Arm/Group | Active First | Active-First Washout | Active-First Then Sham | Active-First-Then-Sham Washout | Active-First Post-Study Monitoring (PSM) Period | Sham First | Sham-First Washout | Sham-First Then Active | Sham-First-Then-Active Washout | Sham-First Post-Study Monitoring (PSM) Period
Number analyzed (Participants) | 41 | 40 | 39 | 39 | 37 | 44 | 40 | 39 | 38 | 37
Points on a Scale | -12.0 (2.3) | -13.1 (2.4) | -16.8 (2.4) | -15.9 (2.0) | -12.1 (2.7) | -6.5 (1.9) | -8.3 (2.0) | -13.8 (2.7) | -13.4 (2.8) | -15.3 (2.6)

3. Primary Outcome: Tinnitus Handicap Inventory (THI)
Description: A 25 item questionnaire which assesses subjective impacts of tinnitus related to quality of life on a 100 point numeric scale. Scores 17 points or higher are considered bothersome tinnitus. The higher scores reflecting greater self-perceived tinnitus handicap. These will be collected weekly during each treatment arm and washout.
  For each of the two arms, Active Then Sham and Sham Then Active, data is presented at the end of each arm phase group, in six week intervals. Thus Active First below is at 6 weeks after baseline, Washout is at 12 weeks, Active First then Sham at 18, and Active First then Sham Washout at 24 and the same pattern for the Sham First group. Values presented are all shown as change from baseline.
Time Frame: Up to 24 weeks
Measure: Mean (Standard Error); unit: Points on a Scale
Arm/Group | Active First | Active-First Washout | Active-First Then Sham | Active-First-Then-Sham Washout | Sham First | Sham-First Washout | Sham-First Then Active | Sham-First-Then-Active Washout
Number analyzed (Participants) | 41 | 40 | 39 | 39 | 44 | 40 | 39 | 38
Points on a Scale | -5.8 (2.1) | -6.4 (1.9) | -8.0 (2.6) | -6.9 (2.0) | -1.6 (1.5) | -2.2 (1.7) | -5.3 (2.8) | -4.6 (2.7)

4. Secondary Outcome: Change in Tinnitus Bandwidth/Spectrum (TinnTester Interactive Software)
Description: Participants are guided through a self-directed computerized assessment software that estimates how similar their tinnitus is to a set of select sounds rated on a 0 - 100 scale where 0 is not similar & 100 is identical. Treatment will relate outcomes to tinnitus bandwidth by these measurements and determine whether the treatment alters bandwidth.
  For each of the two arms, Active Then Sham and Sham Then Active, data is presented at the end of each arm phase group, in six week intervals. Thus Active First below is at 6 weeks after baseline, Washout is at 12 weeks, Active First then Sham at 18, and Active First then Sham Washout at 24 and the same pattern for the Sham First group. Values presented are all shown as change from baseline.
Time Frame: Up to 24 weeks
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Active First | Active-First Washout | Active-First Then Sham | Active-First-Then-Sham Washout | Sham First | Sham-First Washout | Sham-First Then Active | Sham-First-Then-Active Washout
Number analyzed (Participants) | 41 | 40 | 39 | 39 | 44 | 40 | 39 | 38
units on a scale | 7.1 (0.9) | 8.4 (1.0) | 9.5 (1.0) | 10.3 (1.2) | 8.0 (0.9) | 8.5 (1.0) | 10.3 (1.4) | 11.0 (1.5)

5. Secondary Outcome: Changes in Minimum Masking Level (MML)
Description: Determine if the MML for a high-pass 2kHz broadband noise is change in the active treatment arm.
  For each of the two arms, Active Then Sham and Sham Then Active, data is presented at the end of each arm phase group, in six week intervals. Thus Active First below is at 6 weeks after baseline, Washout is at 12 weeks, Active First then Sham at 18, and Active First then Sham Washout at 24 and the same pattern for the Sham First group. Values presented are all shown as change from baseline.
Time Frame: Up to 24 weeks
Measure: Mean (Standard Deviation); unit: dB (sensation level)
Arm/Group | Active First | Active-First Washout | Active-First Then Sham | Active-First-Then-Sham Washout | Sham First | Sham-First Washout | Sham-First Then Active | Sham-First-Then-Active Washout
Number analyzed (Participants) | 41 | 40 | 39 | 39 | 44 | 40 | 39 | 38
dB (sensation level) | -5.1 (2.3) | -1.1 (2.3) | -2.0 (2.9) | 0.2 (2.0) | -2.7 (1.6) | -1.6 (1.5) | 0.0 (2.1) | -0.1 (3.3)

6. Secondary Outcome: Tinnitus Hearing Survey
Description: This is a 10-question survey with a scale from 0 to 4 to determine if active treatment has an effect or interaction with perceived handicap due to hearing loss and sound level tolerance. Categories are comprised of tinnitus, hearing, and sound tolerance. An answer of 0 is no/not a problem, and an answer of 4 is yes/a very big problem. The range for the total score is 0 - 40 with lower numbers meaning fewer hearing problems and higher numbers meaning more tinnitus, or hearing or sound tolerance problems. For each of the two arms, Active Then Sham and Sham Then Active, data is presented at the end of each arm phase group, in six week intervals. Thus Active First below is at 6 weeks after baseline, Washout is at 12 weeks, Active First then Sham at 18, and Active First then Sham Washout at 24 and the same pattern for the Sham First group.
Time Frame: Up to 24 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active First | Active-First Washout | Active-First Then Sham | Active-First-Then-Sham Washout | Sham First | Sham-First Washout | Sham-First Then Active | Sham-First-Then-Active Washout
Number analyzed (Participants) | 41 | 40 | 39 | 39 | 44 | 40 | 39 | 38
score on a scale | -0.7 (0.4) | -1.8 (0.4) | -0.9 (0.5) | -1.4 (0.6) | -0.2 (0.4) | -0.6 (0.5) | -1.3 (0.5) | -1.5 (0.6)

ADVERSE EVENTS:
Time Frame: From screening until end of Post-Study Monitoring (PSM) period up to 36 weeks
Groups:
- Post-Enrollment Through Baseline Measures, Pre-use: all participants prior to use of either device (active or sham)
- Active: All participants while using active device
- Active-Washout Period: All participants in the washout period after active device
- Sham: All participants while on sham device
- Sham-Washout Period: ll participants in the washout period following sham device
- Post-Study Monitoring (PSM): all participants in post-study monitoring
Arm/Group | Post-Enrollment Through Baseline Measures, Pre-use | Active | Active-Washout Period | Sham | Sham-Washout Period | Post-Study Monitoring (PSM)
All-Cause Mortality (participants affected / at risk) | 0/99 | 0/86 | 0/80 | 0/89 | 0/82 | 0/76
Serious Adverse Events (participants affected / at risk) | 0/99 | 0/86 | 0/80 | 0/89 | 0/82 | 0/76
Other Adverse Events (participants affected / at risk) | 3/99 | 19/86 | 9/80 | 16/89 | 12/82 | 1/76
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Post-Enrollment Through Baseline Measures, Pre-use (N=99) | Active (N=86) | Active-Washout Period (N=80) | Sham (N=89) | Sham-Washout Period (N=82) | Post-Study Monitoring (PSM) (N=76)
medical infections (Infections and infestations) | 2 | 9 | 5 | 11 | 11 | 1
ent - head (Ear and labyrinth disorders) | 0 | 7 | 2 | 3 | 1 | 0
worsened tinnitus (Nervous system disorders) | 1 | 4 | 2 | 4 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-02-16): https://cdn.clinicaltrials.gov/large-docs/35/NCT03621735/Prot_SAP_001.pdf
  • Informed Consent Form (2022-02-24): https://cdn.clinicaltrials.gov/large-docs/35/NCT03621735/ICF_000.pdf